CLINICAL TRIAL: NCT04870008
Title: Aesthetic Outcome of Running Cuticular Suture Distance (2mm vs 5mm) From Wound Edge on the Closure of Linear Wounds on the Head and Neck: a Randomized Evaluator Blinded Split Wound Comparative Effective Trial
Brief Title: Aesthetic Outcome of Running Cuticular Suture Distance (2mm vs 5mm)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Daniel Eisen, MD, Professor of Clinical Dermatology, Director of Dermatologic Surgery, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1508837
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Suture; Dermatologic Surgery; Scar; Cosmetic Outcome
MeSH Terms: conditions — Cicatrix | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 mm (Active Comparator): The side of patient's scar that will receive the sutures placed at 2 mm from wound edge.
  Interventions: Procedure: Suture
- 5 mm (Active Comparator): The side of patient's scar that will receive the sutures placed at 5 mm from wound edge.
  Interventions: Procedure: Suture

INTERVENTIONS:
Procedure: Suture — The side of patient's scar that will receive the sutures placed at 2 or 5 mm from wound edge.

SUMMARY:
It is standard teaching that the top layer of sutures should be placed 3-5mm from the wound edge. However, there is lack of data regarding the most optimal placement of sutures from the wound edge for the best cosmetic outcome. The research team wish to determine if sutures placed closer to the wound edge (2mm) or farther from the wound edge (5mm) makes a difference in the cosmetic outcome of the scar.

DETAILED DESCRIPTION:
Sutures are the standard of care in repairing cutaneous wounds. The majority of surgical reconstructions following a Mohs micrographic surgery and standard surgical excisions require two layers of sutures: a deep (subcutaneous) layer and a top (cutaneous) layer. The deep layer dissolves naturally whereas the top layer may necessitate removal if non-absorbable sutures are used. Given the overall lack of evidence in the literature, the choice of suturing technique is largely dependent on the surgeon's preference.

This study aims to investigate whether the distance of simple cuticular suture placement from the wound edge affects wound cosmesis on the head and neck. In other words, we would like to determine which of the following yields a more cosmetically appealing scar: cuticular sutures placed 2 mm from wound edge or cuticular sutures placed 5mm from wound edge.

Although a Dermatologic surgery textbook states that simple cuticular sutures should be placed 3 mm-5 mm from the wound edge1, there have not been any studies to evaluate the optimal distance from wound edge to achieve the most cosmetically appealing scar.

Overall, there is paucity of data regarding the optimal distance of cuticular suture placement from the wound edge to achieve the most cosmetically appealing scar. The research team hope that the study will provide new insight in cutaneous surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the head and neck with predicted primary closure
* Willing to return for follow up visit

Exclusion Criteria:

* Mentally handicapped
* Incarceration
* Under 18 years of age
* Pregnant Women
* Wounds with predicted closure length less than 3 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
The score of two blinded reviewers using the patient observer scar assessment score | 3-12 months
  At the follow-up visit, two blinded observers will record their scores independently using the POSAS (Patient and Observer Scar Assessment Scale) instrument. Each item of the POSAS is rated on a 10-point score. The lowest score is '1', which corresponds to the situation of normal skin (i.e. normal pigmentation, no itching). Score 10 equals the largest difference from normal skin (i.e. the worst imaginable scar or sensation). The total score of both scales can be simply calculated by summing up the scores of each of the six items.
The mean scar width using the trace-to-tape method at the assessment visit | 3-12 months
  The trace-to-tape method is an objective outcome measure for linear postoperative scars. Mean scar width in mm.

SECONDARY OUTCOMES:
Any complications from the treatment | 3-12 months
  Occurrence of any complications including: spitting sutures, dehiscence, infection, necrosis, bleeding, and hematoma

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided